CLINICAL TRIAL: NCT06029257
Title: Effectiveness and Safety of Tildrakizumab in the Treatment of Genital Psoriasis in Austria, Switzerland, and the Czech Republic
Brief Title: A Study of Tildrakizumab in the Treatment of Genital Psoriasis (CZATCH-Genital-PsO)
Status: Recruiting | Type: Observational
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CZATCH-2023
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Genital Psoriasis
Keywords: Psoriasis; Plaque psoriasis; Skin Diseases; Tildrakizumab
MeSH Terms: conditions — Psoriasis; Skin Diseases | interventions — tildrakizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tildrakizumab: Participants who have been prescribed tildrakizumab in the treatment of plaque psoriasis with a manifestation in the genital area according to SmPC in routine clinical practice settings will be observed prospectively for up to 52 weeks.
  Interventions: Drug: Tildrakizumab

INTERVENTIONS:
Drug: Tildrakizumab — As provided in real-world clinical practice.
  Other Names: Ilumetri®

SUMMARY:
The main aim of this study is to check the safety and effectiveness of tildrakizumab regarding the alleviation of symptoms in the genital area after administration according to the summary of product characteristics (SmPC) and to access overall treatment safety and quality of life assessed on multiple scales.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of psoriasis, with significant involvement of genital regions, i.e., sPGA-G greater than or equal to (>=) 3.
* Need for systemic biologic therapy based on the local country specific regulations. Tildrakizumab, in accordance with the SmPC, must be the anti-IL23p19 selected therapy before including the patient in the study.
* Age 18 - 99 years.
* Informed consent in writing in accordance with applicable country regulations
* Patient must have plaque psoriasis affecting a body surface area (BSA) >= 1% in a non-genital area at baseline.
* Patient willing and able to fill out study questionnaires.

Exclusion Criteria:

* Patient appears to be unwilling or unable to comply with the requirements of the study or who, in the opinion of the investigator, should not participate in the study.
* Patient exposed to any experimental treatment in the past 3 months prior to baseline.
* Any condition preventing prescription of Tildrakizumab according to the SmPC, including but not restricted to any contraindication or history of hypersensitivity or intolerance.
* Patient dependent on the investigator, including but not restricted to employees of the study site.
* Previous treatment with Tildrakizumab.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female psoriasis participants with genital symptoms will be observed in this study.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a Static Physician's Global Assessment of Genitalia (sPGA-G) Score of "Clear" (0) or "Almost Clear" (1) | Baseline up to Week 52
  The sPGA-G is a 5-point score ranging from 0 to 4, with a larger score indicating greater severity, based on the physician's assessment of the average thickness, erythema, and scaling of psoriatic genital lesions.
Change From Baseline in Modified Genital Psoriasis Area and Severity Index (mGPASI) Score | Baseline up to Week 52
  mGPASI determines participants psoriasis severity in the genital region at a given time point yielding an overall score of 0 for no psoriasis to 72 for the most severe disease. Scoring index incorporates the degree of erythema (or redness), induration (or thickness), and scaling) of the genital plaques as well as erosion, fissure, and/or ulcer as a product of the genital area involved.

SECONDARY OUTCOMES:
Change From Baseline in Genital Psoriasis Symptoms Scale (GPSS) Score | Baseline, Week 4, 16, 28 and 52
  The GPSS is a self-reported measure where participants were asked to assess each of their psoriasis symptoms (itch, pain, discomfort, stinging, burning, redness, scaling, and cracking) in the genital area and select a number on a scale of 0-10, where 0 represents no symptoms, and 10 represents the worst imaginable. Each symptom assessment were summed to generate a total GPSS score ranging from 0 (no genital psoriasis symptoms) to 80 (worst imaginable genital psoriasis symptoms).
Change From Baseline in Pain, Itch, and Discomfort on Numerical Rating Scales (NRS) for the Genital Region | Baseline, Week 4, 16, 28 and 52
  Genital region is defined as the labia majora (outer lip), labia minora (inner lip), and perineum (area between vagina and anus) for females; penis, scrotum, and perineum (area between the penis and anus) for males. NRS is the simplest and most commonly used scales to indicate the degree of pain, itch, and discomfort. The numerical scale is most commonly 0 to 10, with 0 being "no pain or Itch or discomfort" and 10 being "the worst imaginable pain or Itch or discomfort".
Change From Baseline in the Dermatological Life Quality Index (DLQI) Score | Baseline, Week 4, 16, 28 and 52
  DLQI is a questionnaire which is to evaluate the impact on participant's quality of life due to psoriasis. It is composed of ten items related to symptoms, feelings, daily activities, leisure, working or studying activities, personal relationships and opinions about dermatological treatment. Each item is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life. The higher the score, the more quality of life is impaired.
Change From Baseline in Treatment Satisfaction Questionnaire for Medication (TSQM-9) Score | At Week 28 and 52
  The TSQM-9 is a psychometrically robust and validated instrument to assess participants satisfaction with the treatment they are receiving. It is a self-administered questionnaire that measures participants drug therapy satisfaction considering the last two or three weeks or since the last time the participant took the medication. It consists of 9 items distributed in 3 domains: effectiveness, convenience, and global satisfaction, with scores at each domain ranging from 0 to 100. with higher score indicating higher treatment satisfaction.
Change From Baseline in Genital Psoriasis Sexual Frequency Questionnaire (GenPs-SFQ) Score | Baseline, Week 28 and 52
  The GenPs-SFQ is a participant reported outcome measure to evaluate the impact of genital psoriasis symptoms on sexual frequency. It consists of 2 items that assess the impact of genital psoriasis symptoms on the frequency of sexual activity. Respondents were asked to answer the questions based on their psoriasis symptoms in the genital area. 2 Items assesses how often genital psoriasis symptoms limited the frequency of sexual activity with the following response options: 0 = never, 1 = rarely, 2 = sometimes, 3 = often, 4 = always.
Change from Baseline in Physician's Global Assessment (PGA) Score | Baseline, Week 4, 16, 28 and 52
  The PGA is an instrument used in clinical trials to rate the severity of psoriasis. It is a 5-point scale measurement ranging from 0 to 4, where 0- clear, 1- almost clear, 2- mild, 3- moderate and 4- severe; based on degree of plaque thickening, scaling and erythema.
Change From Baseline in World Health Organisation - 5 Well-Being Index (WHO-5) Score | Baseline, Week 28 and 52
  The WHO-5 consists of 5-items that measure current mental well-being. Each item is rated on 6-point Likert scale, ranging from 0 (at no the time) to 5 (all of the time). The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Universität Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No